CLINICAL TRIAL: NCT04241107
Title: Laparoscopic Versus Transvaginal Approaches in Repair of Uterine Niche: A Randomized Controlled Trial
Acronym: isthmocele
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Abdulrahman Muhammad Rageh, Assistant Lecturer, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Uterine niche repair
Record Dates: First submitted 2020-01-20; First posted 2020-01-27 (Actual); Last update posted 2020-02-05 (Actual); Status verified 2020-02

CONDITIONS: Uterine Niche
Keywords: Cesarean Scar defect

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Laparoscopic approach group(A) (Active Comparator): Uterine niche will be repaired through Laparoscopic approach.
  Interventions: Procedure: Laparoscopic repair of Uterine niche
- Transvaginal approach group(B) (Active Comparator): Uterine niche will be repaired through Transvaginal approach.
  Interventions: Procedure: Transvaginal repair of Uterine niche

INTERVENTIONS:
Procedure: Laparoscopic repair of Uterine niche — Repair of uterine niche through Laparoscopic approach.
  Arms: Laparoscopic approach group(A)
Procedure: Transvaginal repair of Uterine niche — Repair of uterine niche through Transvaginal approach.
  Arms: Transvaginal approach group(B)

SUMMARY:
The treatment of uterine niche ranges from clinical management with expectant or pharmacological treatment, surgical treatment. Approaches for repair include Laparotomy, laparoscopy , hysteroscopy , vaginal. The decision to treat takes into consideration the size of the defect, presence of symptoms, secondary infertility and plans of pregnancy.

All of the approaches have its merits and debates. There is ongoing debate regarding the best surgical approach to managing this condition. To date no randomized controlled trials have been published to settle this debate.

Our study aim is to to evaluate which surgical approach is a preferable option, this study will be conducted to compare the Laparoscopic and transvaginal approaches in several regards, including, operation time, blood loss, perioperative complications, hospital stay length, postoperative increase in residual myometrial thickness during follow-up , clinical efficacy(percentage of patients who subject improvement of symptoms)

ELIGIBILITY:
Inclusion Criteria:

- Patients who have uterine niche (defined as myometrial discontinuity or a hypoechoic triangle in the myometrium of the anterior uterine wall at the site of hysterotomy presented in transvaginal ultrasound or sonohysterography examination in non-pregnant women) ,with one or more previous caesarean section Who are:

1. Symptomatic i.e patients having one or more of the following symptoms:

   1. Postmenstrual spotting (defined as more than 2 days of brownish discharge at the end of menstruation with a total length of menstruation (including spotting) of more than 7 days, or intermenstrual bleeding which starts within 5 days after the end of menstruation. [15]),
   2. Secondary Dysmenorrhea( defined as the pain or discomfort associated with menstruation)
   3. deep dyspareunia(deep genital pain associated with sexual intercourse)
   4. Chronic pelvic pain can be defined as intermittent or constant pain in the lower abdomen or pelvis of a woman of at least 6 months in duration, not occurring exclusively with menstruation or intercourse and not associated with pregnancy.
   5. secondary infertility (defined by the World Health Organization as, -when a woman is unable to bear a child, either due to the inability to become pregnant or the inability to carry a pregnancy to a live birth following either a previous pregnancy or previous ability to carry a pregnancy to a live birth.)
2. Asymptomatic patients with one of the followings:

   the residual myometrial thickness over the niche less than 3 mm previous history of Cesarean Section scar ectopic pregnancy (not managed by resection and repair)
3. who accept to participate the study.

Exclusion Criteria:

1. Asymptomatic patients with residual myometrial thickness more than 3 mm.
2. No previous Cesarean section.
3. If the patients symptoms presented before Cesarean section.
4. Presence of other pathology that explain patient symptoms

   1. sub mucous fibroid
   2. cervical-Endometrial carcinoma
   3. Endometrial hyperplasia
   4. Coagulation defect.
5. Presence of pathology that necessitate laparotomy.
6. Patient who refuse to participate the study.

Ages: 20 Years to 43 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2020-03 (Estimated); Primary Completion 2021-12 (Estimated); Study Completion 2022-03 (Estimated)

PRIMARY OUTCOMES:
Clinical efficacy | 3 month postoperative
  Number of patients who subject clinical improvement of pre-operative symptoms
Post-operative increase in residual myometrial thickness | 3 month postoperative
  difference between pre-operative & post-operative residual myometrial thickness

SECONDARY OUTCOMES:
Duration of operation | baseline( During operation)
  duration from anesthesia till end of operation
Blood loss | baseline( During operation)
  estimated blood loss during operation(towels , suction container)
Intra-operative complication | baseline( During operation)
  complication during the operation

CONTACTS AND LOCATIONS:
Overall Officials: Mahmoud Abdel-Aleem, PhD, Study Chair — Assiut University; Mahmoud zakhera, PhD, Study Chair — Assiut University; Ahmed Abo El Fadle, MD, Study Chair — Assiut University
Locations (1):
- Abdulrahman Muhammad Rageh, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Betran AP, Torloni MR, Zhang JJ, Gulmezoglu AM; WHO Working Group on Caesarean Section. WHO Statement on Caesarean Section Rates. BJOG. 2016 Apr;123(5):667-70. doi: 10.1111/1471-0528.13526. Epub 2015 Jul 22. No abstract available. PMID 26681211
- [Background] Elnakib S, Abdel-Tawab N, Orbay D, Hassanein N. Medical and non-medical reasons for cesarean section delivery in Egypt: a hospital-based retrospective study. BMC Pregnancy Childbirth. 2019 Nov 8;19(1):411. doi: 10.1186/s12884-019-2558-2. PMID 31703638
- [Background] Bij de Vaate AJ, van der Voet LF, Naji O, Witmer M, Veersema S, Brolmann HA, Bourne T, Huirne JA. Prevalence, potential risk factors for development and symptoms related to the presence of uterine niches following Cesarean section: systematic review. Ultrasound Obstet Gynecol. 2014 Apr;43(4):372-82. doi: 10.1002/uog.13199. PMID 23996650
- [Background] Tulandi T, Cohen A. Emerging Manifestations of Cesarean Scar Defect in Reproductive-aged Women. J Minim Invasive Gynecol. 2016 Sep-Oct;23(6):893-902. doi: 10.1016/j.jmig.2016.06.020. Epub 2016 Jul 5. PMID 27393285
- [Background] Vervoort AJ, Uittenbogaard LB, Hehenkamp WJ, Brolmann HA, Mol BW, Huirne JA. Why do niches develop in Caesarean uterine scars? Hypotheses on the aetiology of niche development. Hum Reprod. 2015 Dec;30(12):2695-702. doi: 10.1093/humrep/dev240. Epub 2015 Sep 25. PMID 26409016
- [Background] Sipahi S, Sasaki K, Miller CE. The minimally invasive approach to the symptomatic isthmocele - what does the literature say? A step-by-step primer on laparoscopic isthmocele - excision and repair. Curr Opin Obstet Gynecol. 2017 Aug;29(4):257-265. doi: 10.1097/GCO.0000000000000380. PMID 28598911
- [Background] van der Voet LF, Bij de Vaate AM, Veersema S, Brolmann HA, Huirne JA. Long-term complications of caesarean section. The niche in the scar: a prospective cohort study on niche prevalence and its relation to abnormal uterine bleeding. BJOG. 2014 Jan;121(2):236-44. doi: 10.1111/1471-0528.12542. PMID 24373597
- [Background] Tower AM, Frishman GN. Cesarean scar defects: an underrecognized cause of abnormal uterine bleeding and other gynecologic complications. J Minim Invasive Gynecol. 2013 Sep-Oct;20(5):562-72. doi: 10.1016/j.jmig.2013.03.008. Epub 2013 May 14. PMID 23680518
- [Background] Marotta ML, Donnez J, Squifflet J, Jadoul P, Darii N, Donnez O. Laparoscopic repair of post-cesarean section uterine scar defects diagnosed in nonpregnant women. J Minim Invasive Gynecol. 2013 May-Jun;20(3):386-91. doi: 10.1016/j.jmig.2012.12.006. Epub 2013 Jan 26. PMID 23357466
- [Background] Abacjew-Chmylko A, Wydra DG, Olszewska H. Hysteroscopy in the treatment of uterine cesarean section scar diverticulum: A systematic review. Adv Med Sci. 2017 Sep;62(2):230-239. doi: 10.1016/j.advms.2017.01.004. Epub 2017 May 10. PMID 28500899
- [Background] Ludwin A, Martins WP, Ludwin I. Evaluation of uterine niche by three-dimensional sonohysterography and volumetric quantification: techniques and scoring classification system. Ultrasound Obstet Gynecol. 2019 Jan;53(1):139-143. doi: 10.1002/uog.19181. No abstract available. PMID 30039641
- [Background] Zhang X, Yang M, Wang Q, Chen J, Ding J, Hua K. Prospective evaluation of five methods used to treat cesarean scar defects. Int J Gynaecol Obstet. 2016 Sep;134(3):336-9. doi: 10.1016/j.ijgo.2016.04.011. Epub 2016 Jun 30. PMID 27473332
- [Background] Donnez O, Jadoul P, Squifflet J, Donnez J. Laparoscopic repair of wide and deep uterine scar dehiscence after cesarean section. Fertil Steril. 2008 Apr;89(4):974-80. doi: 10.1016/j.fertnstert.2007.04.024. Epub 2007 Jul 10. PMID 17624346
- [Background] Bij de Vaate AJ, Brolmann HA, van der Voet LF, van der Slikke JW, Veersema S, Huirne JA. Ultrasound evaluation of the Cesarean scar: relation between a niche and postmenstrual spotting. Ultrasound Obstet Gynecol. 2011 Jan;37(1):93-9. doi: 10.1002/uog.8864. PMID 21031351
- See also: Various Types of Niche Imaging by Sonohysterography — http://www.researchgate.net/publication/273145514_Various_Types_of_Niche_Imaging_by_Sonohysterography_A_Pictorial_Review